CLINICAL TRIAL: NCT06565052
Title: The Impact of PReOPerative Exercise and NutritionaL Optimization on Perioperative Outcomes for Patients Undergoing Treatment for Rectal Cancer: The PROPEL Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey A. Meyerhardt, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-384
Record Dates: First submitted 2024-08-16; First posted 2024-08-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer; Colorectal Cancer; Rectal Cancer Stage II; Rectal Cancer Stage III
Keywords: Rectal Cancer; Colorectal Cancer; Rectal Cancer Stage II; Rectal Cancer Stage III
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators blinded to block size
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Prehabilitation Program (Experimental): Participants will be randomized in a 1:1 ratio using a permuted blocked design and stratified by neoadjuvant therapy received. Participants will complete the following:
  * In-clinic baseline visit with assessments
  * Virtual exercise sessions 3 days per week for 4 weeks.
  * IMN supplementation and daily multivitamin starting at 4 weeks of the preoperative phase.
  * Resection surgery per standard of care
  * In-clinic 30 day postoperative visit.
  Interventions: Behavioral: Prehabilitation Program
- Group B: Usual Care (No Intervention): Participants will be randomized in a 1:1 ratio using a permuted blocked design and stratified by neoadjuvant therapy received. Participants will complete the following:
  * In-clinic baseline visit with assessments
  * Resection surgery per standard of care
  * In-clinic 30 day postoperative visit
  * After completion of the study period, participants will be offered exercise equipment with an exercise instruction booklet.

INTERVENTIONS:
Behavioral: Prehabilitation Program — A hybrid-based, prehabilitation regimen comprised of nutritional optimization (multivitamin and protein supplement shake) and virtual, aerobic and resistance exercise sessions with clinical exercise physiologists. Virtual exercise sessions will be performed via a HIPAA-compliant videoconferencing platform or by phone call. Mini-exercise cycle ergometer, dumbbells, and resistance bands will be provided and delivered to participant. Heart rate monitors and wi-fi enable tablet will be provided if needed.
  Arms: Group A: Prehabilitation Program

SUMMARY:
The purpose of this study is to determine the feasibility of a prehabilitation program for participants diagnosed with rectal cancer undergoing neoadjuvant chemotherapy and/or radiation, followed by surgical resection.

The names of the groups in this research study are:

* Group A: Prehabilitation program
* Group B: Usual Care

DETAILED DESCRIPTION:
This is a non-blinded, randomized control trial to determine the feasibility of a hybrid-model, prehabilitation program for participants diagnosed with rectal cancer undergoing neoadjuvant therapy (chemotherapy and/or radiation) before surgical resection. Investigators hope that prehabilitation will result in improved outcomes after surgery.

Participants will be randomized into one of the study groups: Group A: prehabilitation program, or Group B: usual care. Randomization means that a participant is placed into a group by chance.

The research study procedures include screening for eligibility, in-clinic visits, physical exams, exercise training, blood tests, and questionnaires.

It is expected that about 40 participants will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at time of enrollment.
* English-Speaking.
* Diagnosis of clinical stage II-III rectal cancer.
* Planned, ongoing or just completed neoadjuvant treatment, including either 1) chemoradiation, 2) total neoadjuvant therapy (TNT), or 3) chemotherapy only; and anticipated surgical resection to follow.
* Able to understand the study procedures, agree to participate in the study program, and voluntarily provide informed consent.

Exclusion Criteria:

* Distant metastatic disease known at the time of diagnosis.
* Functional incapacity (i.e., incapable of performing exercise testing).
* Comorbid conditions or cognitive/physical impairments that contraindicate exercise.
* Currently undergoing treatment for a secondary primary tumor, in addition to primary rectal cancer.
* Currently enrolled in a separate clinical trial that would prohibit them from performing the tasks instructed in this trial.
* Currently participating in more than 60 minutes of moderate-to-vigorous aerobic exercise per week over the past month. This study targets insufficiently active persons to assess the effect of the described intervention, where additional exercise done regularly will contaminate the intervention effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate | Baseline
  The proportion of eligible individuals that are enrolled to the study. Feasibility of the intervention is defined as an enrollment rate of greater than 10% of approached, eligible participants.

SECONDARY OUTCOMES:
Adherence Rate to the Prehabilitation Program | At post-intervention (approximately Week 4)
  The number of intervention assessments completed by participants in Group A. Feasibility of the intervention is defined as at least 50% of participants adhering to at least 50% of the prescribed assessments of the prehabilitation program.
Completion Rate of Physical Function Testing (Group A) | At post-intervention (approximately Week 4)
  Defined as the number of testing assessments (resting blood pressure, measure of cardiorespiratory fitness, Short Physical Performance Battery, muscular strength, and anthropometric measures) completed by participants.
Completion Rate of Physical Function Testing (Group B) | At post-intervention (approximately Week 4)
  Defined as the number of testing assessments (resting blood pressure, measure of cardiorespiratory fitness, Short Physical Performance Battery, muscular strength, and anthropometric measures) completed by participants.
Completion Rate of Questionnaire Assessments | At baseline and the postoperative visit (approximately Week 9)
  Defined as the number of questionnaires completed by all participants.
Participant Fall Rate (Group A) | At post-intervention (approximately Week 4)
  Defined as the number of falls attributable to the exercise and nutrition components of the intervention.
Participant Fall Rate (Group B) | At post-intervention (approximately Week 4)
  Defined as the number of falls attributable to the exercise and nutrition components of the intervention.
Rate of Hospitalization (Group A) | At post-intervention (approximately Week 4)
  Defined as the number of hospitalizations attributable to the exercise and nutrition components of the intervention.
Rate of Hospitalization (Group B) | At post-intervention (approximately Week 4)
  Defined as the number of hospitalizations attributable to the exercise and nutrition components of the intervention.
Rate of Musculoskeletal Injury (Group A) | At post-intervention (approximately Week 4)
  Defined as the number of musculoskeletal injuries attributable to the exercise and nutrition components of the intervention.
Rate of Musculoskeletal Injury (Group B) | At post-intervention (approximately Week 4)
  Defined as the number of musculoskeletal injuries attributable to the exercise and nutrition components of the intervention.
Change in Resting Blood Pressure from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Assessed by resting blood pressure. The average systolic blood pressure (of two measurements from each arm) will be recorded.
Change in Cardiorespiratory Fitness from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Assessed by VO2peak by a graded maximal (or submaximal if equipment is unavailable) cycle exercise stress test. VO2peak is defined as the highest values of oxygen uptake averaged among every 30-second interval during the test. VO2peak will be reported in both relative (ml·kg-1·min-1) and absolute (L/min) terms.
Change in Short Physical Performance Battery (SPPB) Score from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Assessed by the Short Physical Performance Battery (SPPB) which is comprised of three sections: 1) balance with feet together, semi tandem, and full tandem is held for up to 10 seconds with no support and measure in seconds. Scores are summed for the measure of balance for a range of 0 to 30 seconds; 2) usual gait speed over four meters is timed (seconds); and 3) chair stand where the time(s) to complete five chair sit-to-stands is recorded. Each of the three performance measures is assigned a score ranging from 0 to 4, with 4 indicating highest level of performance and 0 indicating inability to complete test. A summary score ranging from 0 (worst performers) to 12 (best performers) is calculated by adding walking speed, chair stands and balance scores.
Change in Muscle Strength from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  The 1RM (repetition maximum) will be estimated from 10RM muscle strength tests on two exercises: 1) leg press, 2) chest press. 1RM values will be calculated and reported using validated equations.
Change in Height from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Height will be measured using a stadiometer, rounding up to the nearest 0.1 cm
Change in Weight from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Assessed by weight, rounding up to the nearest 0.1 kg.
Change in Waist Circumference from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Waist circumference will be measured, rounding up to the nearest 0.1cm.
Change in Hip Circumference from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Hip circumference will be measured, rounding up to the nearest 0.1cm.
Change in Body Mass Index from Baseline to Post-Intervention | From baseline to post-operative visit (approximately week 9)
  Body composition will be assessed via bioelectrical impedance using a validated device. The device will estimate body fat using an algorithm based on participant age, sex, height, and body weight.
Change in Nutritional Status from Baseline to Post-Surgery (Group A) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the Perioperative Nutrition Score (PONS), a validated screening questionnaire that assists in determining risk of malnutrition in the perioperative setting. This is assessed via 1) Body mass index (BMI), which can be calculated through the participant's anthropomorphic measurements, 2) self-reported unplanned changes in weight or decrease in dietary intake, or 3) preoperative albumin level.
Change in Nutritional Status from Baseline to Post-Surgery (Group B) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the Perioperative Nutrition Score (PONS), a validated screening questionnaire that assists in determining risk of malnutrition in the perioperative setting. This is assessed via 1) Body mass index (BMI), which can be calculated through the participant's anthropomorphic measurements, 2) self-reported unplanned changes in weight or decrease in dietary intake, or 3) preoperative albumin level.
Change in Quality of Life from Baseline to Post-Surgery (Group A) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the European Organization for Research and Treatment of Cancer's (EORTC's) Quality of Life (QOL) core questionnaire (QLQ C-30), a validated, 30-item instrument designed to quantify and measure QOL in cancer participants. Questions are rated on a four point scale from 1 "Not at all" to 4 "Very much. All items have a score range from 0 to 100 points. A higher score represents better function and a higher quality of life.
Change in Quality of Life from Baseline to Post-Surgery (Group B) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the Pittsburgh Sleep Quality Index (PSQI), a 19 question measure of 7 domains of sleep quality and patterns of sleep. The 19 self-rated items are combined to form 7 component scores, each of which has a range of 0 to 3 points with a 0 indicating no difficulty and 3 indicating severe difficulty. The 7 component scores are added to yield a total score with a range of 0 to 21 points. A total score of 5 or greater is indicative of poor sleep quality.
Change in Pittsburgh Sleep Quality Index (PSQI) Score from Baseline to Post-Surgery (Group A) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the Pittsburgh Sleep Quality Index (PSQI), a 19 question measure of 7 domains of sleep quality and patterns of sleep. The 19 self-rated items are combined to form 7 component scores, each of which has a range of 0 to 3 points with a 0 indicating no difficulty and 3 indicating severe difficulty. The 7 component scores are added to yield a total score with a range of 0 to 21 points. A total score of 5 or greater is indicative of poor sleep quality.
Change in PSQI Score from Baseline to Post-Surgery (Group B) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the Pittsburgh Sleep Quality Index (PSQI), a 19 question measure of 7 domains of sleep quality and patterns of sleep. The 19 self-rated items are combined to form 7 component scores, each of which has a range of 0 to 3 points with a 0 indicating no difficulty and 3 indicating severe difficulty. The 7 component scores are added to yield a total score with a range of 0 to 21 points. A total score of 5 or greater is indicative of poor sleep quality.
Change in Clinical Frailty Scale (CFS) Score from Baseline to Post-Surgery (Group A) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the Clinical Frailty Scale (CFS), which consists of 9 questions assessing specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Change in Clinical Frailty Scale (CFS) Score from Baseline to Post-Surgery (Group B) | From baseline to postoperative visit, up to 9 weeks
  Assessed by the Clinical Frailty Scale (CFS), which consists of 9 questions assessing specific domains including comorbidity, function, and cognition to generate a frailty score ranging from 1 (very fit) to 9 (terminally ill).
Length of Hospitalization Post-Surgery (Group A) | 30 Days
  Defined as the number of days of hospitalization post-surgery.
Length of Hospitalization Post-Surgery (Group B) | 30 Days
  Defined as the number of days of hospitalization post-surgery.
Time To Return of Bowel Function Post-Surgery (Group A) | 30 Days
  Defined as the number of days to a return of bowl function post-surgery.
Time To Return of Bowel Function Post-Surgery (Group B) | 30 Days
  Defined as the number of days to a return of bowl function post-surgery.
Discharge Disposition (Group B) | 30 Days
  Defined as participant disposition post-surgery: discharge to home, inpatient rehabilitation facility, or other. Data will be summarized using descriptive statistics.
Discharge Disposition (Group A) | 30 Days
  Defined as participant disposition post-surgery: discharge to home, inpatient rehabilitation facility, or other. Data will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyerhardt, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu